CLINICAL TRIAL: NCT03612089
Title: From Structural to Functional Characteristics of the Lumbar Multifidus in Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Sofie Rummens, MD, KU Leuven
Other Study IDs: s60404
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain group: Individuals with non-specific chronic low back pain
- Healthy control group: Healthy individuals without low back pain

SUMMARY:
To delineate the underlying mechanisms that contribute to chronic low back pain, by extending our knowledge on structural characteristics of the lumbar multifidus muscle using ultrasound muscle imaging, and by examining the association of structural features with functional performance, more precisely proprioceptive control.

ELIGIBILITY:
Inclusion criteria for chronic low back pain group:

* Non-specific low back pain, during 3 or more months, without radicular leg pain
* Modified Low Back Pain Disability Questionnaire > 20%
* Indication for MRI of the lumbar spine
* No contra-indications for MRI
* Informed consent to participate

Inclusion criteria for healthy control group:

* No history of low back pain needing medical treatment or resulting in limited activity level
* Any low back pain in the previous 3 months
* Informed consent to participate

Exclusion criteria for all subjects:

* Pregnancy
* Previous trauma or surgery to spine, abdomen or pelvis
* Structural deformity (e.g. scoliosis)
* Neurological/neuromuscular/systemic disease
* Inability to lie prone for 20 minutes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Leuven and surroudings
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Lumbar multifidus muscle volume measured by 3DfUS | immediately after inclusion in the study
  in patients with chronic low back pain
Lumbar multifidus muscle volume measured by MRI | immediately after inclusion in the study
  in patients with chronic low back pain
Cross-sectional area of the lumbar multifidus | immediately after inclusion in the study
  measured by classic 2D-ultrasound in patients with chronic low back pain and healthy controls
Thickness of the lumbar multifidus | immediately after inclusion in the study
  measured by classic 2D-ultrasound in patients with chronic low back pain and healthy controls
Proprioceptive postural control strategies in patients with low back pain with healthy controls | immediately after inclusion in the study
  Mean center-of-pressure displacement in response to soleus muscle and/or multifidus muscle vibration (60 Hz, 0.5 mm) during upright standing on two support surfaces.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No